CLINICAL TRIAL: NCT03987126
Title: Use of Novel Human Milk Prebiotics to Improve the Quality of Life for Spinal Cord Injury Patients With Bowel and Bladder Dysfunction
Brief Title: Prebiotics for Spinal Cord Injury Patients With Bowel and Bladder Dysfunction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: The W. Garfield Weston Foundation (Unknown); St. Joseph's Health Care London (Other); Parkwood Hospital, London, Ontario (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 6170
Record Dates: First submitted 2019-06-04; First posted 2019-06-14 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Spinal Cord Injuries; Neurogenic Bowel; Bladder Dysfunction
MeSH Terms: conditions — Spinal Cord Injuries; Neurogenic Bowel | interventions — Health Maintenance Organizations

STUDY DESIGN:
Intervention Model Description: One placebo arm and one active treatment arm, participants will be assigned to each arm equally based on their Neurogenic Bowel Dysfunction score.
Who Masked: Participant, Care Provider, Investigator
Masking Description: No other parties will be masked for the study. A part of the study will be open label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Human Milk Oligosaccharide (HMO) (Active Comparator): 10 g sachet, self-administered for 3 months.
  2'-O-fucosyllactose and lacto-N-neotetraose, novel human milk oligosaccharide (HMO) sugars have already been shown to very specifically modulate intestinal bacteria, namely the beneficially viewed bifidobacteria, in clinical studies in adults. Modulating bifidobacteria increases the levels of specific short chain fatty acids (SCFAs), such as butyrate, propionate and acetate.These SCFAs have been shown to stimulate colonic sodium and fluid absorption and exert proliferative effects on the colonocyte in experimental animal studies since the 1990s (Scheppach 1994). Therefore, increasing their levels would lead to an improvement in intestinal motility, as has been summarised previously (Koh 2016)
  Interventions: Dietary Supplement: Human Milk Oligosaccharides (HMO)
- Placebo (Placebo Comparator): 10 g sachet, self-administered for 3 months.
  Placebo sachets are identical to the HMO sachets in color, taste, smell, size and shape
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Human Milk Oligosaccharides (HMO) — Sachet containing 10 grams of HMO
  Arms: Human Milk Oligosaccharide (HMO)
Other: Placebo — Sachet manufactured to mimic 10g of HMO
  Other Names: Placebo for HMO
  Arms: Placebo

SUMMARY:
An investigator initiated pilot study: two arm, double blind, placebo controlled, randomized, group of approximately 60 patients with spinal cord injury, and who have evidence of neurogenic bladder. Patients will be treated with human milk oligosaccharide (HMO) versus placebo over 12 weeks from start of the investigational medication date (approximately 3 months) to test whether HMO can improve bowel motility in neurogenic bowel and bladder patients. Patients in the placebo arm of the study will be offered participation in the open label portion of the study immediately after their part in the control group is completed, they will receive HMO for 12 weeks. HMO sachets will be administered to determine the safety and efficacy of HMO relative to placebo in improving quality of life of neurogenic bowel and bladder patients by improving bowel motility and function.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) is a life changing neurologic diagnosis that affects multiple body systems. Urinary tract infections (UTIs) are almost a universal complication of SCI with bladder dysfunction, and a significant cause of morbidity in those with SCI. Recurrent UTIs requires multiple courses of antibiotic therapy, increasing the incidence of multidrug-resistant bacteria. While curative antibiotic therapy is transiently effective, recurrences are frequent and bladder colonization is inevitable after SCI because of an impaired ability to empty the bladder. Meta-analysis of SCI and UTI have shown there is no evidence to support the use of prophylactic antibiotics. Although the exact mechanism of action is not fully understood, nearly all UTIs are caused by bacteria from the bowel. Therefore, addressing the impaired bowel function in SCI patients would not only improve this debilitating condition but also reduce UTI's and the need for antibiotic therapy.

Since prebiotics are metabolised by bacteria in the colon and their by-products promote intestinal peristalsis and can relieve constipation, they could represent an effective option to treat bowel dysfunction in SCI patients. The study's aim is to improve bowel motility in SCI patients with neurogenic bowel impairments by using 2'-O-fucosyllactose and lacto-N-neotetraose, novel human milk oligosaccharide (HMO) sugars that have already been shown to very specifically modulate intestinal bacteria. In the bowel, the HMO would induce an increase in bifidobacteria, which would further produce short chain fatty acids such that stimulate bowel motility and other beneficially regarded bacteria.

The Principal Investigator/Sponsor will test this potential in a pilot clinical study with a HMO mix that has shown to promote bifidobacteria (Ellison 2016). These HMO compounds are structurally different from the less pure, plant-or bovine dairy-based prebiotics that are currently used in other human applications, and are safe, well tolerated, food grade substances. They have been shown to soften the stools in healthy adults and reduce constipation; therefore, it is expected they will positively impact the quality of life of neurogenic bowel and bladder patients by improving bowel motility, and also reducing the associated co-morbidity of recurrent urinary tract infections. The study will collect data on a sample of up to 60 patients with SCI and neurogenic bowel dysfunction scores of >13.

The Principal Investigator/Sponsor will assess the HMO's effects on the quality of life, intestinal bacterial composition, bowel motility, and associated co-morbidities such as urinary tract infections (UTIs). In the longer term this is expected to reduce UTI occurrence due to reduced pathogen loading; as a consequence, reduce antibiotic use and levels of drug resistant bacteria.If the study If successful, the results outlining its significance could be forwarded to the senior management team at the recruiting hospital to be considered as a potential management tool in the care of patients with SCI.

This study will assess faecal and urine samples at four time points for microbiome and other analyses at baseline, 4 weeks, 8 weeks (approximately 2 months) and 12 weeks (approximately 3 months) from the date of starting the study product. Prior to commencing their treatment, and at weeks 8 and 12, the research coordinator (blinded to the randomisation) will assess patients using various bowel, bladder and quality of life questionnaires during clinic visits, at home or by telephone interview.

The type, level, and completeness of injury will be documented, and the type of bowel and bladder dysfunction (upper or lower motor neuron) will be classified and, if necessary, updated at each in-person visit. Each participant will be provided with instructions and study schedule.

Protocol compliance will be tested through product count and interviews at each follow-up visit. Side effects will be assessed using standardized case report forms at each visit. Study visits may be in person or over the phone. Participants will be encouraged to report any events they may experience directly to the coordinator.

Participants who withdraw consent to continue treatments, will be encouraged to undergo the planned assessments. Withdrawal at the request of investigators or medical personnel may include, but are not limited to:

1. Symptoms are deemed to be potentially related to the study product
2. New diagnosis of exclusion criteria;
3. Unacceptable side effects;
4. Death

Estimated time to complete recruitment: Averaging 53 weeks, approximately 12 months

ELIGIBILITY:
Inclusion Criteria:

* 18 years old
* SCI of at least 3 months duration
* Neurogenic bowel dysfunction scores of >10 OR 4 or less bowel movements per week, OR requires a suppository to have a bowel movement

Exclusion Criteria:

* Pregnancy
* Inability to understand and respond to the provided questionnaires
* Carcinomas during the last 5 years
* Bowel surgery
* Crohn ́s disease or other bowel conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Bowel motility | 12 weeks
  Improvement of 25-30% in our study population in the neurogenic bowel function of our intervention study group after treatment, will be measured by the Neurogenic Bowel dysfunction score. Neurogenic Bowel Dysfunction score will be measured by a symptom-based questionnaire that scores 10 variables to attain a total score between 0 and 47. It includes frequency of bowel movements, time of defecation, evacuation and incontinence.
Neurogenic bowel dysfunction score (NBD) | 12 weeks
  The change in this assessment from baseline to end of study will help determine the improvement in bowel motility. It is a symptom-based questionnaire that scores 10 variables to attain a total score between 0 and 47. It includes frequency of bowel movements, time of defecation, evacuation and incontinence.
Change in method of bowel assistance | 12 weeks
  Medications required, home remedies used, other methods of assistance will be recorded in a study questionnaire.
Duration of bowel routine | 12 weeks
  Measured by the NBD questionnaire.
Episodes of incontinence | 12 weeks
  Will be measured in time between bowel movements by the NBD questionnaire.
Frequency of bowel movements per week | 12 weeks
  Will be measured by the NBD questionnaire.

SECONDARY OUTCOMES:
Microbiome changes from baseline to end of study | 12 weeks
  Changes in the entire bacterial community from baseline to end of study will be assessed in the lab from faecal and urine samples collected by the participant. The microbes may vary by participant and the study will be looking at which ones present themselves in each case. Of particular interest may be the Enterobacteriaceae like Escherichia coli that cause UTI. Units of measure via culture are colony forming units per g (cfu/g).
Changes in pain | 12 weeks
  A modified International Spinal Cord Injury Pain Basic Dataset version 2.0 questionnaire will be used. The first part of the questionnaire is a scale that ranges from 1-10, with 1 stating their pain is not interfering with their daily activities, and 10 stating extreme interference. The second part is a table that lists different areas of the body and has the participant check off whether they feel pain in the right, middle, or left side of each body area. Pain type will be assessed by the referring clinician and documented in a study CRF.
Change in sleep | 12 weeks
  will be documented in the International Spinal Cord Injury Pain Basic Dataset v2.0 questionnaire. The question scales from 1 - 10, 1 stating that pain has had no interference with the participant getting a good night's sleep, and 10 stating major interference.
Change in mood | 12 weeks
  will be documented in the International Spinal Cord Injury Pain Basic Dataset v2.0 questionnaire. The answer will be measured in a scale from 1-10, 1 stating that pain has had no interference with their mood, and 10 stating major interference.
Quality of Life Measures survey | 12 weeks
  a general quality of life measures survey will be included in the study. The QOLS is scored by adding up the score on each item to yield a total score for the instrument. The cale includes 16 questions, each question can be answered from a range of 1-7 (1 being very unhappy, 7 being very happy) Scores can range from 16 to 112.
Number of participants reporting unexpected adverse events | 12 weeks
  Adverse events will be recorded through case report forms and reported to the principal investigator. Side effects will be assessed using standardized case report forms at each visit. Participants are encouraged to contact the coordinator to report any concerns.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy P Burton, PhD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- Parkwood Institute, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Taweel WA, Seyam R. Neurogenic bladder in spinal cord injury patients. Res Rep Urol. 2015 Jun 10;7:85-99. doi: 10.2147/RRU.S29644. eCollection 2015. PMID 26090342
- [Background] Krogh K, Christensen P, Sabroe S, Laurberg S. Neurogenic bowel dysfunction score. Spinal Cord. 2006 Oct;44(10):625-31. doi: 10.1038/sj.sc.3101887. Epub 2005 Dec 13. PMID 16344850
- [Background] Christensen P, Bazzocchi G, Coggrave M, Abel R, Hultling C, Krogh K, Media S, Laurberg S. A randomized, controlled trial of transanal irrigation versus conservative bowel management in spinal cord-injured patients. Gastroenterology. 2006 Sep;131(3):738-47. doi: 10.1053/j.gastro.2006.06.004. PMID 16952543
- [Background] Christensen P, Bazzocchi G, Coggrave M, Abel R, Hulting C, Krogh K, Media S, Laurberg S. Outcome of transanal irrigation for bowel dysfunction in patients with spinal cord injury. J Spinal Cord Med. 2008;31(5):560-7. doi: 10.1080/10790268.2008.11754571. PMID 19086714
- [Background] Tulsky DS, Kisala PA, Tate DG, Spungen AM, Kirshblum SC. Development and psychometric characteristics of the SCI-QOL Bladder Management Difficulties and Bowel Management Difficulties item banks and short forms and the SCI-QOL Bladder Complications scale. J Spinal Cord Med. 2015 May;38(3):288-302. doi: 10.1179/2045772315Y.0000000030. PMID 26010964
- [Background] Elison E, Vigsnaes LK, Rindom Krogsgaard L, Rasmussen J, Sorensen N, McConnell B, Hennet T, Sommer MO, Bytzer P. Oral supplementation of healthy adults with 2'-O-fucosyllactose and lacto-N-neotetraose is well tolerated and shifts the intestinal microbiota. Br J Nutr. 2016 Oct;116(8):1356-1368. doi: 10.1017/S0007114516003354. Epub 2016 Oct 10. PMID 27719686
- [Background] Koh A, De Vadder F, Kovatcheva-Datchary P, Backhed F. From Dietary Fiber to Host Physiology: Short-Chain Fatty Acids as Key Bacterial Metabolites. Cell. 2016 Jun 2;165(6):1332-1345. doi: 10.1016/j.cell.2016.05.041. PMID 27259147
- [Background] Al KF, Bisanz JE, Gloor GB, Reid G, Burton JP. Evaluation of sampling and storage procedures on preserving the community structure of stool microbiota: A simple at-home toilet-paper collection method. J Microbiol Methods. 2018 Jan;144:117-121. doi: 10.1016/j.mimet.2017.11.014. Epub 2017 Nov 16. PMID 29155236
- [Background] Bao Y, Al KF, Chanyi RM, Whiteside S, Dewar M, Razvi H, Reid G, Burton JP. Questions and challenges associated with studying the microbiome of the urinary tract. Ann Transl Med. 2017 Jan;5(2):33. doi: 10.21037/atm.2016.12.14. PMID 28217698
- [Background] Reid G, Burton JP. Urinary incontinence: Making sense of the urinary microbiota in clinical urology. Nat Rev Urol. 2016 Oct;13(10):567-8. doi: 10.1038/nrurol.2016.182. Epub 2016 Sep 20. No abstract available. PMID 27644934
- [Background] Whiteside SA, Razvi H, Dave S, Reid G, Burton JP. The microbiome of the urinary tract--a role beyond infection. Nat Rev Urol. 2015 Feb;12(2):81-90. doi: 10.1038/nrurol.2014.361. Epub 2015 Jan 20. PMID 25600098
- [Background] Scheppach W. Effects of short chain fatty acids on gut morphology and function. Gut. 1994 Jan;35(1 Suppl):S35-8. doi: 10.1136/gut.35.1_suppl.s35. PMID 8125387
- See also: The first canadian national atlas of Spinal Cord Injury Rehabilitation from a collaborative community of practice to provide the best care to individuals living with the consequences of spinal cord injury. — https://rickhanseninstitute.org/e-scan-atlas